CLINICAL TRIAL: NCT03743064
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Anamorelin HCl for the Treatment of Malignancy Associated Weight Loss and Anorexia in Adult Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study to Evaluate the Efficacy and Safety of Anamorelin HCl for the Treatment of Malignancy Associated Weight Loss and Anorexia in Adult Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAM-17-21; 2018-002927-40 (EudraCT Number)
Record Dates: First submitted 2018-11-14; First posted 2018-11-15 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Cachexia; Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Cachexia; Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Multicenter Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This was a double-blind study. The blinding of the study drugs was guaranteed by the use of anamorelin HCl film-coated tablets and matching placebo tablets. Patients were randomized using the Interactive Web Response System (IWRS). Any unblinding of the study treatment was performed using the IWRS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100 mg anamorelin HCl (Experimental): 100 mg anamorelin HCl (administered as film-coated tablets in fasted condition) was to be taken orally once daily for a total of 24 weeks
  Interventions: Drug: anamorelin HCl
- Placebo (Placebo Comparator): Placebo (administered as matching placebo tablets in fasted condition) was to be taken orally once daily for a total of 24 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: anamorelin HCl — 100 mg anamorelin HCl (administered as 100 mg tablets in the fasted condition)
  Arms: 100 mg anamorelin HCl
Drug: Placebo Oral Tablet — Placebo (administered as matching placebo tablets in the fasted condition)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial was to compare the efficacy and safety of anamorelin HCl (the investigational drug) to that of placebo (tablet with no drug) in patients with advanced non-small cell lung cancer and cachexia (cancer-related weight loss). The main question it aimed to answer was as follows: Do patients who receive anamorelin HCl gain more body weight and show more improvement in anorexia symptoms than those who receive placebo.

Approximately 316 patients were to be enrolled in the study. Of these patients, an equal number were to be assigned to each treatment group (anamorelin HCl or placebo). Participants were to take their assigned study drug by mouth once daily for a total of 24 weeks. During this treatment period, the patients were to visit the clinical study site every 3 weeks for health and other study-related assessments. Two weeks after the last treatment, patients were to receive a follow-up phone call.

DETAILED DESCRIPTION:
The study was a multicenter, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy and safety of anamorelin HCl. It was planned that approximately 316 patients with advanced NSCLC with cachexia were to be randomized 1:1 to anamorelin HCl 100 mg or placebo (158 patients per treatment group). The study treatment was to be taken orally once daily for a total of 24 weeks. Patients were instructed to take the study drug at least 1 hour before their first meal of the day.

Central randomization was stratified by line of systemic anti-cancer treatment (first line vs second line vs third line or higher), by type of anti-cancer therapy (immunotherapy vs non-immunotherapy), and by baseline score of 5 IASS (≤10 vs >10). Patients who had never received anti-cancer treatment prior to entering the study but who met all eligibility criteria were eligible to enter the study and were assigned to receive first line treatment in the Interactive Web Response System (IWRS).

Patients were to visit the site every 3 weeks for the study Treatment Period of 24 weeks. A follow-up telephone visit was to be scheduled at Week 26. Thus, patients were enrolled in the study for a maximum duration of 27 weeks (including a 1-week Screening Period, a 24-week Treatment Period, and a 2-week Follow-up Period). Each patient was scheduled to have a total of 10 planned visits plus 1 telephone contact for the Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Female or male ≥18 years of age
3. Documented histologic or cytologic diagnosis of American Joint Committee on Cancer (AJCC) Stage III or IV NSCLC. Stage III patient must have unresectable disease
4. Body mass index < 20 kg/m2 with involuntary weight loss of >2% within 6 months prior to screening
5. Ongoing problems with appetite/eating associated with the underlying cancer, as determined by having score of ≤ 17 points on the 5-item Anorexia Symptom Scale and ≤ 37 points on the 12-item FAACT A/CS
6. Patient receiving or not receiving systemic anti-cancer treatment at the time of screening are eligible to participate. Systemic anti-cancer treatment includes first, second, third treatment line with chemotherapy/radiation therapy, immunotherapy or targeted therapy.

   Patient not receiving systemic anti-cancer treatment is eligible if:
   1. Not planning to receive anti-cancer treatment and/or at least 14 days must be elapsed from the completion of prior treatment at the day of screening, in case underwent previous cycle OR
   2. Planning to receive anti-cancer treatment within 14 days from randomization and/or at least 14 days must be elapsed from the completion of prior treatment at the day of screening, in case underwent previous cycle OR
   3. Patient on palliative care treatment
7. ECOG performance status 0,1 or 2 at screening
8. AST (SGOT) and ALT (SGPT) ≤ 3 x ULN or if hepatic metastases are present ≤ 5 x ULN
9. Adequate renal function, defined as creatinine ≤2 ULN, or calculated creatinine clearance >30 ml/minute
10. Female patient shall be: a) of non-childbearing potential or b) of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test within 24 hours prior to first dose of investigational product.

    Notes:
    1. Female patient of non-childbearing potential are defined as being in post-menopausal state since at least 1 year; or having documented surgical sterilization or hysterectomy at least 3 months before study participation.
    2. Reliable contraceptive measures include implants, injectables, combined oral contraceptives, intrauterine devices, vasectomized partner or complete (long term) sexual abstinence.
11. The patient must be willing and able to comply with the protocol tests and procedures All inclusion criteria will be checked at screening visit (Visit 1).

Exclusion Criteria:

1. Patient with other forms of lung cancer (e.g., small cell, neuroendocrine tumors)
2. Woman who is pregnant or breast-feeding
3. Reversible causes of reduced food intake, as determined by the Investigator. These causes may include but are not limited to:

   1. NCI CTCAE Grade 3 or 4 oral mucositis,
   2. NCI CTCAE Grade 3 or 4 GI disorders [nausea, vomiting, diarrhea, and constipation],
   3. mechanical obstructions making patient unable to eat, or
   4. severe depression
4. Patient undergoing major surgery (central venous access placement and tumor biopsies are not considered major surgery) within 4 weeks prior to randomization. Patient must be well recovered from acute effects of surgery prior to screening. Patient should not have plans to undergo major surgical procedures during the treatment period
5. Patient currently taking androgenic compounds (including but not limited to testosterone, testosterone-like agents, oxandrolone, megestrol acetate, corticosteroids, olanzapine, mirtazapine (however, long-term use of mirtazapine for depression for at least four weeks prior to screening is allowed), dronabinol or marijuana (cannabis) or any other prescription medication or off-label products intended to increase appetite or treat unintentional weight loss
6. Patient with pleural effusion requiring thoracentesis, pericardial effusion requiring drainage, edema or evidence of ascites
7. Patient with uncontrolled or significant cardiovascular disease, including:

   1. History of myocardial infarction within the past 3 months
   2. A-V block of second or third degree (may be eligible if currently have a pacemaker)
   3. Unstable angina
   4. Congestive heart failure within the past 3 months, if defined as NYHA class III-IV
   5. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, Wolff-Parkinson-White (WPW) syndrome, or torsade de pointes)
   6. Uncontrolled hypertension (blood pressure >150 mm Hg systolic and >95 mm Hg diastolic)
   7. Heart rate < 50 beats per minute on pre-entry electrocardiogram and patient is symptomatic
8. Patient on drugs that may prolong the PR or QRS interval durations, such as any of the antiarrhythmic medications Class I (Fast sodium (Na) channel blockers)
9. Patient unable to readily swallow oral tablets
10. Patient with severe gastrointestinal disease (including esophagitis, gastritis, malabsorption)
11. Patient with history of gastrectomy
12. Patient with uncontrolled diabetes mellitus or unmonitored diabetes mellitus
13. Patient with cachexia caused by other reasons, as determined by the investigator such as:

    1. Severe COPD requiring use of home O2,
    2. New York Heart Association (NYHA) class III-IV heart failure
    3. AIDS
    4. Uncontrolled thyroid disease
14. Patient receiving strong CYP3A4 inhibitors within 14 days of randomization
15. Patient currently receiving tube feedings or parenteral nutrition (either total or partial).
16. Current excessive alcohol or illicit drug use
17. Any condition, including the presence of laboratory abnormalities, which in the Investigator's opinion, places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
18. Enrollment in a previous study with anamorelin HCl
19. Patient actively receiving a concurrent investigational agent, or having received an investigational agent within 28 days of Day 1 All exclusion criteria will be checked at screening visit (Visit 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (19):
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - CBCC Global Research Inc, Bakersfield, California
  - Compassionate Care Research Group, Inc., at Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Marin Cancer Care, Greenbrae, California
  - Smilow Cancer Hospital at Yale-New Haven, Waterbury, Connecticut
  - Bond & Steele Clinic P.A., Winter Haven, Florida
  - Presence Infusion Care, Skokie, Illinois
  - Siouxland Regional Cancer Center dba June E.Nylen Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New Jersey Hematology Oncology Associates Inc, Brick, New Jersey
  - Hunterdon Hematology Oncology LLC, Flemington, New Jersey
  - Hematology Oncology Center at Nyack Hospital, Nyack, New York
  - University of Rochester, Medical Center, Rochester, New York
  - Duke Cancer Center, Durham, North Carolina
  - Toledo Clinic Cancer Center-Toledo, Toledo, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Calvary Central Districts Hospital, Elizabeth Vale, South Australia
  - Flinders Medical Centre, Bedford Park
  - St Vincent's Hospital Melbourne, Fitzroy
  - Barwon Health, The McKellar Centre, North Geelong
  - The Royal Melbourne Hospital, Parkville
  - Gold Coast University Hospital, Southport
- Belgium (5):
  - Jules Bordet Institut, Brussels
  - Saint Luc University Hospital, Brussels
  - Charleroi Grand Hospital (GHDC), Charleroi
  - University Hospital Antwerp (UZA), Edegem
  - General Hospital Delta, Roeselare
- Croatia (3):
  - General Hospital Pula, Pula
  - University Hospital Center Split, Split
  - University Hospital Center Zagreb, Zagreb
- Poland (7):
  - Wladyslaw Bieganski Regional Specialist Hospital, Clinical Oncology Department, Grudziądz
  - "VEGAMED" Non-Public Healthcare Facility, Katowice
  - MSF Institute Ltd. Santa Familia Medical Institute, Lodz
  - MED - POLONIA Ltd., Poznan
  - Specialist Hospital in Prabuty sp. z o.o. [limited liability company], Department of Pulmonology, Prabuty
  - Maria Skfodowska-Curie Institute of Oncology, Department of Lung and Thoracic Cancers, Warsaw
  - Mazovian Oncology Hospital, Oncology Outpatient Clinic, Wieliszew
- Romania (7):
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Medical Oncology Department, Cluj-Napoca, Cluj
  - "Sf. Nectarie" Oncology Center, Medical Oncology Department, Craiova, Dolj
  - SC Oncopremium Team SRL, Medical Oncology Department, Baia Mare, Maramureş
  - Topmed Medical Center, Medical Oncology Department, Târgu Mureş, Murers
  - Sf. Ioan cel Nou Country Emergency Hospital, Oncology Department, Suceava, Suceava
  - S.C. Oncomed SRL, Medical Oncology Department, Timișoara, Timiș County
  - Alexandru Trestioreanu Institute of Oncology, Bucharest
- Russia (10):
  - Republican Clinical Oncology Center, Kazan'
  - Pyatigorsk Interdistric Oncology Center, Pyatigorsk
  - Oncology Center of Moskovskiy District, Saint Petersburg
  - AV Medical Group, Saint Petersburg
  - Palliative Care Center Devita, Saint Petersburg
  - City Clinical Oncology Center, Saint Petersburg
  - Samara Regional Clinical Oncology Center, Samara
  - Ogaryov Mordovia National Research State University, Republican Oncology Center, Saransk
  - Oncology Center #2, Sochi
  - Volgograd Regional Clinical Oncology Center, Volgograd
- Ukraine (8):
  - Publ Non- Profit Ent. under Kharkiv Reg. Council, Kharkiv, Kharkiev Region
  - Communal Non-Profit Enterprise "Regional Center of Oncology", Kharkiv, Kharkiev
  - Medical Center "VERUM" Limited Liability Company, Kyiv, Kyviv
  - Public Entreprise "Poltava Regional Clinical Oncology Center under Poltava Regional Council", Poltava, Poltava Oblast
  - Medical Center "MEDICAL PLAZA" of the Limited Liability Company "EKODNIPRO", Dnipro
  - Private Enterprise "First Private Clinic", Kyiv
  - Public Non-Profit Enterprise 'Ternopil Regional Clinical Oncology Center'' under Temopil Regional Council, Ternopil
  - Medical Center of Limited Liability Company "ONCOLIFE", Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at a total of 49 study sites in Australia (2 sites), Belgium (2 sites), Croatia (3 sites), Germany (3 sites), Poland (5 sites), Romania (7 sites), Russia (10 sites), Ukraine (8 sites), and USA (9 sites). First Patient Enrollment (date of randomization) was on 06MAY2019.
Pre-assignment Details: The protocol had pre-defined criteria regarding health and medication requirements to begin study drug administration, and if the patient's status for these requirements changed between screening and Study Day 1, treatment could not be initiated.
Period: Overall Study
Arm/Group | 100 mg Anamorelin HCl | Placebo
Started (Randomized) | 154 | 164
Treated | 154 | 164
Completed | 83 | 90
Not Completed | 71 | 74
Not completed — Adverse Event | 7 | 9
Not completed — Death | 25 | 28
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 28 | 25
Not completed — Physician Decision | 2 | 4
Not completed — Reported as "Other" in Clinical Study Report | 6 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Set included all randomized patients and was analyzed as per planned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg Anamorelin HCl | Placebo | Total
Number analyzed (Participants) | 154 | 164 | 318
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (8.49) | 63.6 (9.73) | 63.8 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 50 | 92
  Male | 112 | 114 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 146 | 156 | 302
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 4 | 8
  Black or African American | 0 | 2 | 2
  White | 148 | 157 | 305
  Other | 0 | 1 | 1
  Multiple | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 58 | 59 | 117
  Belgium | 2 | 3 | 5
  United States | 8 | 8 | 16
  Ukraine | 38 | 34 | 72
  Poland | 11 | 19 | 30
  Australia | 1 | 3 | 4
  Croatia | 5 | 5 | 10
  Russia | 27 | 29 | 56
  Germany | 4 | 4 | 8
Height [Mean (Standard Deviation); unit: cm] | 171.03 (8.690) | 169.96 (9.164) | 170.48 (8.940)
Weight [Mean (Standard Deviation); unit: kg] | 54.09 (7.029) | 52.84 (7.925) | 53.44 (7.519)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.38 (1.328) | 18.16 (1.579) | 18.27 (1.465)
Chemotherapy Line [Count of Participants; unit: Participants]
  First Line | 104 | 104 | 208
  Second Line | 36 | 39 | 75
  Third Line | 14 | 21 | 35
Anti-cancer Treatment [Count of Participants; unit: Participants]
  Immunotherapy | 39 | 46 | 85
  Non-immunotherapy | 115 | 118 | 233
5-IASS Score [Count of Participants; unit: Participants] — FAACT-A/CS (Functional Assessment Anorexia Cachexia Therapy) is a 12-item measure of patients' perceptions of anorexia/cachexia symptoms and concerns. From this questionnaire, the 5-item section referring to anorexia symptoms (i.e., "good appetite," "interest in food drops," "food tastes unpleasant," "get full quickly," and "difficulty eating rich/heavy foods") was used to assess 5-IASS. The range of possible scores is 0-20. Higher scores indicate lower levels of symptom burden.
  Participants
    ≤10 | 102 | 107 | 209
    >10 | 52 | 57 | 109
NSCLC stage at study entry [Count of Participants; unit: Participants] — American Joint Committee on Cancer (AJCC) staging for non-small cell lung cancer (NSCLC): The earliest stage of NSCLC is stage 0 (also called carcinoma in situ, or CIS). Other stages range from I through IV. As a rule, the lower the number, the less the cancer has spread. A higher number, such as stage IV, means cancer has spread more. And within a stage, an earlier letter (or number) means a lower stage.
  Participants
    IIIA | 2 | 1 | 3
    IIIB | 30 | 19 | 49
    IV | 122 | 143 | 265
    Missing | 0 | 1 | 1
Body weight change within 6 months prior to screening [Mean (Standard Deviation); unit: percent change] | -10.03 (6.177) | -10.86 (6.612) | -10.46 (6.408)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Body Weight Over 12 Weeks
Description: This co-primary efficacy endpoint was mean change from baseline in body weight (kg) over 12 weeks in the anamorelin HCl group versus placebo group. Mean change was computed as sum of the changes from baseline over 12 weeks by the time of the last assessment (either week 12 or before in case of death), and then divided by the number of assessments (observed or imputed) from baseline up to the time of the last assessment.
Time Frame: Mean change from baseline over 12 weeks.
Population: The Intent-to-Treat (ITT) Set included all randomized patients and was analyzed as per planned treatment.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | 100 mg Anamorelin HCl | Placebo
Number analyzed (Participants) | 154 | 164
kg | 1.822 (0.263) | 0.538 (0.250)
Statistical Analysis 1: Comparison: 100 mg Anamorelin HCl vs Placebo; To declare anamorelin superior to placebo, both co-primary endpoints had to be significant. The null hypothesis for mean change in body weight from baseline over 12 weeks (H0w) and the corresponding alternative hypothesis (H1w) were: H0w: MWa = MWp H1w: MWa ≠ MWp Where MWa is the mean change in body weight from baseline over 12 weeks for the anamorelin arm and MWp is the mean change in body weight from baseline over 12 weeks for the placebo arm; Test type: Superiority — The Multiple Imputation process (N=100) was performed leading to least squares mean (LSM) and standard error (SE) estimates using the ANOVA model (including treatment group and the 3 stratification factors at randomization as categorical covariates). The estimates were pooled using Rubin rule, with corresponding p-value for difference between treatment groups. The 95% confidence interval (CI) was calculated for each treatment group and for the pooled difference between the groups; p < 0.0001, ANOVA; Mean Difference (Final Values) = 1.284, 95% CI 2-sided [0.718 to 1.851], Standard Error of Mean 0.289

2. Primary Outcome: Mean Change From Baseline in 5-item Anorexia Symptom Subscale (5-IASS) Over 12 Weeks
Description: This co-primary efficacy endpoint was mean change from baseline in 5-IASS (points) over 12 weeks in the anamorelin HCl group versus placebo group. Mean change was computed as sum of the changes from baseline over 12 weeks by the time of the last assessment (either week 12 or before in case of death), and then divided by the number of assessments (observed or imputed) from baseline up to the time of the last assessment.
  FAACT-A/CS (Functional Assessment Anorexia Cachexia Therapy) is a 12-item measure of patients' perceptions of anorexia/cachexia symptoms and concerns. From this questionnaire, the 5-item section referring to anorexia symptoms (i.e., "good appetite," "interest in food drops," "food tastes unpleasant," "get full quickly," and "difficulty eating rich/heavy foods") was used to assess 5-IASS. The range of possible scores is 0-20. Higher scores indicate lower levels of symptom burden.
Time Frame: Mean change from baseline over 12 weeks.
Population: The ITT Set included all randomized patients and was analyzed as per planned treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 100 mg Anamorelin HCl | Placebo
Number analyzed (Participants) | 154 | 164
score on a scale | 3.432 (0.360) | 3.291 (0.342)
Statistical Analysis 1: Comparison: 100 mg Anamorelin HCl vs Placebo; To declare anamorelin superior to the placebo, both co-primary endpoints had to be significant. The null hypothesis for mean change from baseline over 12 weeks in patient 5-IASS (H0A) and the corresponding alternative (H1A) were: H0A: MAa = MAp; H1A: MAa ≠ MAp Where MAa is the mean change from baseline over 12 weeks in 5-IASS for the anamorelin arm and MAp is the mean change from baseline over 12 weeks in 5-IASS for the placebo arm; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7241, ANOVA; Mean Difference (Final Values) = 0.141, 95% CI 2-sided [-0.641 to 0.923], Standard Error of Mean 0.399

3. Secondary Outcome: Duration in Treatment Benefit (Weeks) From Baseline Over 12 Weeks in Body Weight (≥0 kg)
Description: The duration of treatment benefit over 12 weeks was measured as the period, or the sum of the periods, over 12 weeks (or less in case of death), in which the patient observed a change from baseline in body weight of ≥0 kg.
Time Frame: Duration of treatment benefit from baseline over 12 weeks.
Population: The ITT Set included all randomized patients and was analyzed as per planned treatment.
Measure: Least Squares Mean (Standard Error); unit: weeks
Arm/Group | 100 mg Anamorelin HCl | Placebo
Number analyzed (Participants) | 154 | 164
weeks | 8.859 (0.525) | 6.778 (0.496)
Statistical Analysis 1: Comparison: 100 mg Anamorelin HCl vs Placebo; Test type: Superiority — All secondary endpoints were analyzed using the same statistical model and multiple imputation approach as for the co-primary efficacy endpoints; p = 0.0003, ANOVA; Mean Difference (Final Values) = 2.081, 95% CI 2-sided [0.946 to 3.216], Standard Error of Mean 0.579

4. Secondary Outcome: Duration in Treatment Benefit (Weeks) From Baseline Over 12 Weeks in Body Weight (≥1.5 kg)
Description: The duration of treatment benefit over 12 weeks was measured as the period, or the sum of the periods, over 12 weeks (or less in case of death), in which the patient observed a change from baseline in body weight of ≥1.5 kg.
Time Frame: Duration of treatment benefit from baseline over 12 weeks.
Population: The ITT Set included all randomized patients and was analyzed as per planned treatment.
Measure: Least Squares Mean (Standard Error); unit: weeks
Arm/Group | 100 mg Anamorelin HCl | Placebo
Number analyzed (Participants) | 154 | 164
weeks | 5.490 (0.431) | 3.087 (0.409)
Statistical Analysis 1: Comparison: 100 mg Anamorelin HCl vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, ANOVA; Mean Difference (Final Values) = 2.404, 95% CI 2-sided [1.471 to 3.337], Standard Error of Mean 0.476

5. Secondary Outcome: Duration of Treatment Benefit (Weeks) From Baseline Over 12 Weeks in 5-IASS (≥0 Points)
Description: The duration of treatment benefit over 12 weeks was measured as the period, or the sum of the periods, over 12 weeks (or less in case of death), in which the patient observed a change from baseline in 5- IASS of ≥0 points.
Time Frame: Duration of treatment benefit from baseline over 12 weeks.
Population: The ITT Set included all randomized patients and was analyzed as per planned treatment.
Measure: Least Squares Mean (Standard Error); unit: weeks
Arm/Group | 100 mg Anamorelin HCl | Placebo
Number analyzed (Participants) | 154 | 164
weeks | 9.470 (0.392) | 8.842 (0.370)
Statistical Analysis 1: Comparison: 100 mg Anamorelin HCl vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1443, ANOVA; Mean Difference (Final Values) = 0.629, 95% CI 2-sided [-0.215 to 1.472], Standard Error of Mean 0.431

6. Secondary Outcome: Duration of Treatment Benefit (Weeks) From Baseline Over 12 Weeks in 5-IASS (≥3 Points)
Description: The duration of treatment benefit over 12 weeks was measured as the period, or the sum of the periods, over 12 weeks (or less in case of death), in which the patient observed a change from baseline in 5- IASS of ≥3 points.
Time Frame: Duration of treatment benefit from baseline over 12 weeks.
Population: The ITT Set included all randomized patients and was analyzed as per planned treatment.
Measure: Least Squares Mean (Standard Error); unit: weeks
Arm/Group | 100 mg Anamorelin HCl | Placebo
Number analyzed (Participants) | 154 | 164
weeks | 5.143 (0.410) | 4.992 (0.387)
Statistical Analysis 1: Comparison: 100 mg Anamorelin HCl vs Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.7376, ANOVA; Mean Difference (Final Values) = 0.151, 95% CI 2-sided [-0.734 to 1.036], Standard Error of Mean 0.452

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of Informed Consent signature through Day 183 (+3) days post study drug administration on Day 1.
Description: The "Serious Adverse Events" and "Other (Not Including Serious) Adverse Events" tables include only treatment-emergent AEs.
Arm/Group | 100 mg Anamorelin HCl | Placebo
All-Cause Mortality (participants affected / at risk) | 25/154 | 28/164
Serious Adverse Events (participants affected / at risk) | 44/154 | 46/164
Other Adverse Events (participants affected / at risk) | 114/154 | 127/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Anamorelin HCl (N=154) | Placebo (N=164)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18) | 19 (19)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleura effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disability (Social circumstances) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (2)
Death (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Anamorelin HCl (N=154) | Placebo (N=164)
Asthenia (General disorders) | 19 (24) | 22 (26)
Chest Pain (General disorders) | 13 (14) | 9 (10)
Fatigue (General disorders) | 7 (7) | 2 (2)
Oedema Peripheral (General disorders) | 7 (9) | 5 (8)
Nausea (Gastrointestinal disorders) | 18 (28) | 12 (16)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 6 (6)
Vomiting (Gastrointestinal disorders) | 6 (8) | 6 (9)
Abdominal Pain (Gastrointestinal disorders) | 5 (6) | 4 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (5) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 28 (33) | 38 (53)
Neutropenia (Blood and lymphatic system disorders) | 10 (10) | 6 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (11) | 4 (6)
Leukopenia (Blood and lymphatic system disorders) | 6 (6) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Sinus Tachycardia (Cardiac disorders) | 7 (7) | 13 (15)
Atrial Fibrillation (Cardiac disorders) | 6 (7) | 5 (6)
Sinus Bradycardia (Cardiac disorders) | 3 (3) | 4 (4)
Ventricular Extrasystoles (Cardiac disorders) | 3 (3) | 4 (5)
Atrioventricular Block (Cardiac disorders) | 2 (2) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5)
Dizziness (Nervous system disorders) | 12 (12) | 5 (5)
Headache (Nervous system disorders) | 9 (9) | 5 (6)
Blood Creatinine Increased (Investigations) | 5 (6) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (7) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (5) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (14)
Nasopharyngitis (Infections and infestations) | 5 (6) | 1 (1)
Corona Virus Infection (Infections and infestations) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the sole right to first publication of the study data, which would be a multi-center publication. Investigators may publish the Study Data they obtained if they follow the conditions provided in the protocol. These include, but are not limited to: the multi-center publication has occurred; the Sponsor is given 60 days to review the document and possibly 60 more days to obtain Intellectual Property protections; and all Confidential Information is deleted, as requested by Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03743064/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03743064/SAP_001.pdf